CLINICAL TRIAL: NCT00439322
Title: Post Traumatic Stress Disorder Among VA Ambulatory Care Patients
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 96-030
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: PTSD
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Posttraumatic stress disorder (PTSD) occurs in response to an extreme traumatic stressor. It is estimated that as many as 1 million VA patients who were exposed to combat may have PTSD. VA patients with PTSD recently have been designated as a �Special Emphasis� population for which health care resources are allocated at approximately 14 times those allocated to patients without such chronic, complex, and intensive health care needs (i.e., �Basic Care� groups). Despite recognition of its substantial impact upon VA resources, the extent and means by which PTSD affects health and health care use remain unclear. This study seeks to enhance understanding of both the extent and means by which PTSD affects the health and the health care use of patients in VA ambulatory care. To meet this goal, we build on an ongoing HSR&D project, the Veterans Health Study (VHS), a prospective longitudinal study of 2,425 VA ambulatory care patients.

DETAILED DESCRIPTION:
Background:

Posttraumatic stress disorder (PTSD) occurs in response to an extreme traumatic stressor. It is estimated that as many as 1 million VA patients who were exposed to combat may have PTSD. VA patients with PTSD recently have been designated as a �Special Emphasis� population for which health care resources are allocated at approximately 14 times those allocated to patients without such chronic, complex, and intensive health care needs (i.e., �Basic Care� groups). Despite recognition of its substantial impact upon VA resources, the extent and means by which PTSD affects health and health care use remain unclear. This study seeks to enhance understanding of both the extent and means by which PTSD affects the health and the health care use of patients in VA ambulatory care. To meet this goal, we build on an ongoing HSR&D project, the Veterans Health Study (VHS), a prospective longitudinal study of 2,425 VA ambulatory care patients.

Objectives:

Posttraumatic stress disorder (PTSD) often afflicts victims of traumatic events such as combat. Growing evidence suggests that PTSD is related to poorer health status and to increased use of health care services. However, the extent of these effects and the means by which they occur remain unclear. The goal of this study is to enhance our understanding of both the extent and means by which PTSD affects the health and the health care use of patients in VA ambulatory care. To meet this goal, we built on an HSR&D service-directed project, the Veterans Health Study (VHS), a prospective longitudinal study of 2,425 male VA ambulatory care patients.

Methods:

This project consisted of two phases. In Phase 1, we conducted clinical interviews (CAPS) assessing PTSD with 474 patients participating in the VHS at 1-year follow-up (T12). This phase validated a brief 17-item self-report PTSD screening measure (PCL-C) against a PTSD clinical interview diagnosis. We used the results of this validation study to estimate the prevalence of PTSD in VA primary care, and to propose the use of a brief measure (PRIME-MD) as a screen for PTSD in primary care. In Phase 2, we used the PCL-C to examine the impact of PTSD on health status and health care use. We tested the hypotheses that (a) PTSD has a direct effect on health status that is independent of the effects of comorbid medical conditions, depression, and alcohol use, and (b) that controlling for comorbid medical conditions, depression and alcohol use, PTSD has both a direct effect and an indirect effect (through health status) on health care utilization. These hypotheses are being tested using structural equation methods. If, as hypothesized, PTSD exerts direct and indirect effects on health services use, then both quality of care and efficiencies in health services delivery can be improved through appropriate detection, referral, and treatment of PTSD among patients in VA ambulatory care.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Veterans enrolled at hospitals where study is implemented.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 473 (Estimated)
Dates: Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avron Spiro, PhD MS, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA; Cheryl S Hankin, PhD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA; Cheryl S Hankin, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

REFERENCES:
- [Result] Hankin CS, Skinner KM, Sullivan LM, Miller DR, Frayne S, Tripp TJ. Prevalence of depressive and alcohol abuse symptoms among women VA outpatients who report experiencing sexual assault while in the military. J Trauma Stress. 1999 Oct;12(4):601-12. doi: 10.1023/A:1024760900213. PMID 10646179
- [Result] Chatterjee S, Rath ME, Spiro A 3rd, Eisen S, Sloan KL, Rosen AK. Gender differences in veterans health administration mental health service use: effects of age and psychiatric diagnosis. Womens Health Issues. 2009 May-Jun;19(3):176-84. doi: 10.1016/j.whi.2009.03.002. PMID 19447322